CLINICAL TRIAL: NCT00866918
Title: Risk Adapted Treatment of Newly Diagnosed Childhood Acute Promyelocytic Leukemia (APL) Using Arsenic Trioxide (Trisenox® ) During Consolidation
Brief Title: Combination Chemotherapy in Treating Young Patients With Newly Diagnosed Acute Promyelocytic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAML0631; NCI-2011-01904 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000637184; AAML0631 (Other: Children's Oncology Group); AAML0631 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Childhood Acute Promyelocytic Leukemia With PML-RARA; Myeloid Neoplasm
MeSH Terms: interventions — Arsenic Trioxide; arsenous acid; Cytarabine; Idarubicin; Mercaptopurine; azathiopurine; Methotrexate; merphos; Mitoxantrone; Tretinoin

ARMS (2):
- Arm I (standard risk, combination chemotherapy) (Experimental): See Detailed Description
  Interventions: Drug: Arsenic Trioxide; Drug: Cytarabine; Other: Diagnostic Laboratory Biomarker Analysis; Drug: Idarubicin; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Mitoxantrone Hydrochloride; Drug: Tretinoin
- Arm II (high risk, combination chemotherapy) (Experimental): See Detailed Description.
  Interventions: Drug: Arsenic Trioxide; Drug: Cytarabine; Other: Diagnostic Laboratory Biomarker Analysis; Drug: Idarubicin; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Mitoxantrone Hydrochloride; Drug: Tretinoin

INTERVENTIONS:
Drug: Arsenic Trioxide — Given IV
  Other Names: Arsenic (III) Oxide; Arsenic Sesquioxide; Arsenous Acid; Arsenous Acid Anhydride; Arsenous Oxide; ATO; Trisenox; White Arsenic
Drug: Cytarabine — Given IT or IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Other: Diagnostic Laboratory Biomarker Analysis — Correlative studies
Drug: Idarubicin — Given IV
  Other Names: 4-Demethoxydaunomycin; 4-Demethoxydaunorubicin; 4-DMDR
Drug: Mercaptopurine — Given orally
  Other Names: 3H-Purine-6-thiol; 6 MP; 6 Thiohypoxanthine; 6 Thiopurine; 6-Mercaptopurine; 6-Mercaptopurine Monohydrate; 6-MP; 6-Purinethiol; 6-Thiopurine; 6-Thioxopurine; 6H-Purine-6-thione, 1,7-dihydro- (9CI); 7-Mercapto-1,3,4,6-tetrazaindene; Alti-Mercaptopurine; Azathiopurine; Bw 57-323H; Flocofil; Ismipur; Leukerin; Leupurin; Mercaleukim; Mercaleukin; Mercaptina; Mercaptopurinum; Mercapurin; Mern; NCI-C04886; Puri-Nethol; Purimethol; Purine, 6-mercapto-; Purine-6-thiol (8CI); Purine-6-thiol, monohydrate; Purinethiol; Purinethol; U-4748; WR-2785
Drug: Methotrexate — Given orally
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Drug: Mitoxantrone Hydrochloride — Given IV
  Other Names: CL 232315; DHAD; DHAQ; Dihydroxyanthracenedione Dihydrochloride; Mitoxantrone Dihydrochloride; Mitoxantroni Hydrochloridum; Mitozantrone Hydrochloride; Mitroxone; Neotalem; Novantrone; Onkotrone; Pralifan
Drug: Tretinoin — Given orally
  Other Names: 2,4,6,8-Nonatetraenoic acid, 3, 7-dimethyl-9-(2,6,6-trimethyl-1-cyclohexen-1-yl)-, (all-E)-; Aberel; Airol; Aknoten; all trans-Retinoic acid; All-trans Retinoic Acid; All-trans Vitamin A Acid; all-trans-Retinoic acid; all-trans-Vitamin A acid; ATRA; Avita; beta-Retinoic Acid; Cordes Vas; Dermairol; Epi-Aberel; Eudyna; Renova; Retin-A; Retin-A MICRO; Retin-A-Micro; Retinoic Acid; Retisol-A; Ro 5488; Stieva-A; Stieva-A Forte; Trans Retinoic Acid; Trans Vitamin A Acid; trans-Retinoic Acid; Tretinoinum; Vesanoid; Vitamin A Acid; Vitamin A acid, all-trans-; Vitinoin

SUMMARY:
This phase III trial is studying combination chemotherapy to see how well it works in treating young patients with newly diagnosed acute promyelocytic leukemia. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To decrease the total anthracycline dose from the best current published results in standard risk childhood acute promyelocytic leukemia (APL) while still maintaining a comparable event-free survival (EFS).

SECONDARY OBJECTIVES:

I. To assign treatment based on risk stratification by white blood cell count (WBC) at diagnosis.

II. To estimate the induction failure rate, toxic death rate, disease-free survival rate and overall survival rate in both standard and high risk APL patients.

III. To monitor for cardiotoxicity in an idarubicin/mitoxantrone based regimen. IV. To document the toxicity of a traditional chemotherapy/all-trans retinoic acid (ATRA) (tretinoin) based regimen combined with arsenic trioxide therapy.

V. To study the relationship of Fms-like tyrosine kinase 3 (FLT3) mutations to clinical features and outcome in APL.

VI. To study risk factors for pseudotumor cerebri in APL. VII. To study the relationship of early progenitor cell involvement to treatment failure in FLT3 positive APL.

VIII. To compare the EFS of children enrolled on AAML0631 with the EFS of children enrolled on C9710 who were between the ages of 2 and 21 and did not receive arsenic trioxide.

IX. To estimate the proportion of patients who carry a cryptic t(15;17), i.e., those who are positive for a promyelocytes.(PML)-retinoic acid receptor alpha (RARA) fusion transcript by polymerase chain reaction (PCR) analysis but have normal chromosomes.

X. To estimate the proportion of patients with variant RARA partners. XI. To compare the outcome of patients with only a t(15;17) with that of patients who carry a t(15;17) and other chromosomal abnormalities.

OUTLINE: This is a multicenter study. Patients are assigned to 1 of 2 arms based on risk factor (standard-risk [WBC less than 10,000/mm^3] or high-risk [WBC 10,000/mm^3 or higher]).

ARM I (STANDARD-RISK):

INDUCTION THERAPY: Patients receive tretinoin orally (PO) twice daily (BID) on days 1-30 and idarubicin intravenously (IV) over 15 minutes once on days 3, 5, and 7.

CONSOLIDATION THERAPY:

CONSOLIDATION 1: Patients receive arsenic trioxide IV over 2 hours on days 1-5, 8-12, 15-19, 22-26, and 29-33 and tretinoin PO BID on days 1-14. Treatment repeats every 5 weeks for 2 courses, followed by a 2-week break, and then treatment repeats for 2 more courses. Beginning 1 week later or when blood counts recover, patients proceed to consolidation 2.

CONSOLIDATION 2: Patients receive cytarabine intrathecally (IT) on day 1, tretinoin PO BID on days 1-14, high-dose cytarabine IV over 3 hours every 12 hours on days 1-3, and mitoxantrone hydrochloride IV over 15-30 minutes once on days 3 and 4. Patients proceed to consolidation 3 1 week later or when blood counts recover.

CONSOLIDATION 3: Patients receive cytarabine IT on day 1, tretinoin PO BID on days 1-14, and idarubicin IV over 15 minutes once daily on days 1, 3, and 5. High-risk patients and those standard-risk patients who are positive for minimal residual disease by real-time quantitative (RQ)-PCR receive consolidation 4 one week later or when blood counts recover. All other standard-risk patients proceed to maintenance therapy.

MAINTENANCE THERAPY: Patients receive cytarabine IT on day 1 (course 1 only), tretinoin PO BID on days 1-14, mercaptopurine PO once daily (QD) on days 1-84, methotrexate PO once on days 1, 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78. Treatment repeats every 12 weeks for 9 courses.

ARM II (HIGH-RISK):

INDUCTION THERAPY: Patients receive tretinoin PO BID on days 1-30 and idarubicin IV over 15 minutes once on days 1, 3, and 5. Patients proceed to consolidation therapy one week later or when blood counts recover.

CONSOLIDATION THERAPY: Patients receive consolidation 1, 2, and 3 as in Arm I.

CONSOLIDATION 4: Patients receive cytarabine IT on day 1, tretinoin PO BID on days 1-14, high-dose cytarabine IV over 3 hours every 12 hours on days 1-3, and idarubicin IV over 15 minutes once on day 4. Patients who demonstrate molecular complete remission (CR) and remain in hematological CR proceed to maintenance therapy 1 week later or when blood counts recover.

MAINTENANCE THERAPY: Patients receive maintenance therapy as in Arm I.

After completion of study treatment, patients are followed every month for 1 year, every 3 months for 2 years, every 6 months for 2 years, and then annually for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be newly diagnosed with a clinical diagnosis of acute promyelocytic leukemia initially by morphology (bone marrow or peripheral blood); bone marrow is highly preferred but in cases where marrow cannot be obtained at diagnosis, peripheral blood will be accepted; APL is considered a hematological emergency and treatment should be initiated as quickly as possible without waiting for molecular or cytogenetic/fluorescence in situ hybridization (FISH) confirmation; for patients who are unable to begin receiving ATRA in a timely manner following a presumed diagnosis of APL, consideration should be given to initiating ATRA and proceeding with treatment outside of the AAML0631 protocol; if the RQ-PCR results are known at the time of study enrollment, the patient must demonstrate PML-RARA and/or RARA-PML transcripts by RQ-PCR to be eligible; patients without evidence of APL by bone marrow or peripheral blood morphology but with isolated myeloid sarcoma (myeloblastoma; chloroma, including leukemia cutis) are eligible provided that the t(15;17) translocation is documented on either marrow or tumor tissue by cytogenetics, FISH, or PCR prior to study enrollment; in this situation, touch preps from the tumor site can be evaluated by FISH with PML-RARA probes; NOTE: A lumbar puncture is not required to be enrolled on study; if the diagnosis of APL is known or suspected, extreme caution must be exercised in performing a lumbar puncture during active coagulopathy; in addition a computed tomography (CT) or magnetic resonance imaging (MRI) should be considered to rule out the possibility of an associated chloroma if central nervous system (CNS) disease is suspected or proven; if CNS disease is documented, patients are still eligible
* No minimal performance status criteria
* The patient must not have received systemic definitive treatment for APL or other suspected leukemia, including cytotoxic chemotherapy, retinoids, or arsenic; prior therapy with corticosteroids, hydroxyurea, or leukopheresis will not exclude the patient; if a patient received intrathecal cytarabine prior to the diagnosis of APL being known, the patient will still be eligible as long as they meet all other eligibility requirements

Exclusion Criteria:

* Pregnant women or nursing mothers are excluded; treatment under this protocol would expose an unborn child to significant risks; patients should not be pregnant or plan to become pregnant while on treatment; women and men of reproductive potential should agree to use an effective means of birth control; there is an extremely high risk of fetal malformation if pregnancy occurs while on ATRA in any amount even for short periods
* Patients with a pre-existing prolonged QT Syndrome will not be eligible for this protocol due to the use of arsenic trioxide which can prolong the QT interval

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 106 (Actual)
Dates: Start 2009-03-09 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John J Gregory, Principal Investigator — Children's Oncology Group
Locations (121):
- United States (112):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Harbor-University of California at Los Angeles Medical Center, Torrance, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Connecticut, Farmington, Connecticut
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Memorial Health System, Fort Myers, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Oncology Group, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (8):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec
- San Jorge Children's Hospital, San Juan, Puerto Rico

REFERENCES:
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Risk: WBC<10,000/MicroLiter
- High Risk: WBC>=10,000/MicroLiter
Period: Overall Study
Arm/Group | Standard Risk | High Risk
Started | 69 | 39
Completed | 53 | 27
Not Completed | 16 | 12
Not completed — Death | 1 | 5
Not completed — Lack of Efficacy | 1 | 1
Not completed — Physician Decision | 10 | 2
Not completed — Ineligible | 2 | 4
Not completed — Inevaluable- RQPCR negative at diagnosi | 1 | 0
Not completed — Secondary malignancy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Risk | High Risk | Total
Number analyzed (Participants) | 69 | 39 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 68 | 38 | 106
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Days] | 4915.25 (1627.27) | 4921.33 (1747.04) | 4917.44 (1663.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 25 | 62
  Male | 32 | 14 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 7 | 23
  Not Hispanic or Latino | 51 | 31 | 82
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 4 | 12
  White | 52 | 30 | 82
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 2 | 9
Region of Enrollment [Number; unit: participants]
  Canada | 2 | 2 | 4
  United States | 67 | 37 | 104

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS)
Description: EFS - time from study entry until failure to achieve complete remission during consolidation, relapse, or death. For further clarification see definitions provided in the protocol.
Time Frame: At 3 years from study entry
Population: Ineligible and inevaluable patients are excluded from analyses of EFS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Standard Risk | High Risk
Number analyzed (Participants) | 66 | 35
Percentage of participants | 95.4 [86.3 to 98.5] | 82.9 [65.8 to 91.9]

2. Secondary Outcome: Hematologic Remission Rate
Description: Proportion of patients in hematologic remission at end of consolidation, course 1 are reported.
Time Frame: End of consolidation, course 1: up to 5 months
Population: Patients who were ineligible (n=6), inevaluable (n=1), or who electively withdrew during Induction (n=4) were excluded.
Measure: Number; unit: Proportion of participants
Arm/Group | Standard Risk | High Risk
Number analyzed (Participants) | 63 | 34
Proportion of participants | 1.0000 | 0.8824

3. Secondary Outcome: Hematologic, Molecular, and Cytogenetic Remission Rate
Description: Proportion of patients in hematologic, molecular, and cytogenetic remission at end of consolidation, course 3 and 4 are reported. Patients were determined to be in remission by all three criteria.
Time Frame: End of consolidation, course 3; up to 7 months (for Standard Risk) or end of consolidation, course 4; up to 9 months (for High Risk)
Population: Patients who were ineligible (n=6), inevaluable (n=1), or who electively withdrew during Induction (n=4) were excluded.
Measure: Number; unit: Proportion of participants
Arm/Group | Standard Risk | High Risk
Number analyzed (Participants) | 63 | 34
Proportion of participants | 0.8095 | 0.5882

4. Secondary Outcome: Overall Survival (OS)
Description: OS - time from study entry to death.
Time Frame: At 3 years from study entry
Population: Ineligible and inevaluable patients are excluded from analyses of OS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Standard Risk | High Risk
Number analyzed (Participants) | 66 | 35
Percentage of participants | 98.4 [89.6 to 99.8] | 85.7 [69.0 to 93.8]

ADVERSE EVENTS:
Description: Patients who were study ineligible (n=6) or inevaluable (n=1, RQ-PCR negative at diagnosis) were excluded from number at risk in the Serious and Other Adverse event data tables.
Arm/Group | Standard Risk | High Risk
Serious Adverse Events (participants affected / at risk) | 17/66 | 14/35
Other Adverse Events (participants affected / at risk) | 61/66 | 33/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Risk (N=66) | High Risk (N=35)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 — Adeers submitted
Acidosis (Metabolism and nutrition disorders) | 0 | 1 — Adeers submitted
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 2 — Adeers submitted
Alanine aminotransferase increased (Investigations) | 1 | 1 — Adeers submitted
Anorexia (Metabolism and nutrition disorders) | 1 | 0 — Adeers submitted
Aspartate aminotransferase increased (Investigations) | 1 | 1 — Adeers submitted
Asystole (Cardiac disorders) | 0 | 1 — Adeers submitted
Blood bilirubin increased (Investigations) | 0 | 1 — Adeers submitted
Bronchial infection (Infections and infestations) | 1 | 0 — Adeers submitted
Catheter related infection (Infections and infestations) | 2 | 3 — Adeers submitted
Dehydration (Metabolism and nutrition disorders) | 1 | 1 — Adeers submitted
Depression (Psychiatric disorders) | 0 | 1 — Adeers submitted
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 — Adeers submitted
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Adeers submitted
Endocarditis infective (Infections and infestations) | 0 | 1 — Adeers submitted
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 1 — Adeers submitted
Fever (General disorders) | 0 | 1 — Adeers submitted
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 — Adeers submitted
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 — Adeers submitted
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 — Adeers submitted
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 — Adeers submitted
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 — Adeers submitted
Hypotension (Vascular disorders) | 3 | 1 — Adeers submitted
Infections and infestations - Other, specify (Infections and infestations) | 4 | 3 — Adeers submitted
INR increased (Investigations) | 0 | 1 — Adeers submitted
Multi-organ failure (General disorders) | 0 | 2 — Adeers submitted
Nausea (Gastrointestinal disorders) | 1 | 1 — Adeers submitted
Neutrophil count decreased (Investigations) | 0 | 1 — Adeers submitted
Pain (General disorders) | 1 | 0 — Adeers submitted
Platelet count decreased (Investigations) | 0 | 1 — Adeers submitted
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 — Adeers submitted
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 — Adeers submitted
Sepsis (Infections and infestations) | 2 | 3 — Adeers submitted
Sinus tachycardia (Cardiac disorders) | 0 | 1 — Adeers submitted
Skin infection (Infections and infestations) | 1 | 0 — Adeers submitted
Syncope (Nervous system disorders) | 0 | 1 — Adeers submitted
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — Adeers submitted
Urinary tract infection (Infections and infestations) | 1 | 0 — Adeers submitted
Vomiting (Gastrointestinal disorders) | 1 | 1 — Adeers submitted
White blood cell decreased (Investigations) | 0 | 1 — Adeers submitted
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Risk (N=66) | High Risk (N=35)
Abdominal pain (Gastrointestinal disorders) | 3 | 4 — Adeers not subm
Acidosis (Metabolism and nutrition disorders) | 0 | 1 — Adeers not subm
Activated partial thromboplastin time prolonged (Investigations) | 2 | 2 — Adeers not subm
Acute kidney injury (Renal and urinary disorders) | 1 | 2 — Adeers not subm
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 1 — Adeers not subm
Agitation (Psychiatric disorders) | 1 | 0 — Adeers not subm
Alanine aminotransferase increased (Investigations) | 14 | 7 — Adeers not subm
Alkaline phosphatase increased (Investigations) | 0 | 2 — Adeers not subm
Allergic reaction (Immune system disorders) | 1 | 0 — Adeers not subm
Anal pain (Gastrointestinal disorders) | 1 | 1 — Adeers not subm
Anemia (Blood and lymphatic system disorders) | 1 | 0 — Adeers not subm
Anorectal infection (Infections and infestations) | 1 | 0 — Adeers not subm
Anorexia (Metabolism and nutrition disorders) | 5 | 5 — Adeers not subm
Appendicitis (Infections and infestations) | 0 | 1 — Adeers not subm
Appendicitis perforated (Infections and infestations) | 0 | 1 — Adeers not subm
Arachnoiditis (Nervous system disorders) | 1 | 0 — Adeers not subm
Ascites (Gastrointestinal disorders) | 1 | 0 — Adeers not subm
Aspartate aminotransferase increased (Investigations) | 8 | 2 — Adeers not subm
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Adeers not subm
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 — Adeers not subm
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 2 | 0 — Adeers not subm
Blood bilirubin increased (Investigations) | 5 | 2 — Adeers not subm
Bone infection (Infections and infestations) | 1 | 0 — Adeers not subm
Bronchial infection (Infections and infestations) | 1 | 0 — Adeers not subm
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 | 0 — Adeers not subm
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Adeers not subm
Cardiac disorders - Other, specify (Cardiac disorders) | 1 | 2 — Adeers not subm
Catheter related infection (Infections and infestations) | 7 | 4 — Adeers not subm
Cholecystitis (Hepatobiliary disorders) | 0 | 1 — Adeers not subm
Colitis (Gastrointestinal disorders) | 1 | 1 — Adeers not subm
Constipation (Gastrointestinal disorders) | 2 | 0 — Adeers not subm
Creatinine increased (Investigations) | 0 | 1 — Adeers not subm
Dehydration (Metabolism and nutrition disorders) | 2 | 1 — Adeers not subm
Depression (Psychiatric disorders) | 1 | 0 — Adeers not subm
Diarrhea (Gastrointestinal disorders) | 3 | 2 — Adeers not subm
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 4 | 3 — Adeers not subm
Dysarthria (Nervous system disorders) | 1 | 0 — Adeers not subm
Dysphagia (Gastrointestinal disorders) | 1 | 0 — Adeers not subm
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 — Adeers not subm
Ear pain (Ear and labyrinth disorders) | 1 | 0 — Adeers not subm
Electrocardiogram QT corrected interval prolonged (Investigations) | 16 | 6 — Adeers not subm
Enterocolitis (Gastrointestinal disorders) | 1 | 0 — Adeers not subm
Enterocolitis infectious (Infections and infestations) | 3 | 1 — Adeers not subm
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 — Adeers not subm
Esophageal infection (Infections and infestations) | 1 | 0 — Adeers not subm
Esophageal pain (Gastrointestinal disorders) | 0 | 1 — Adeers not subm
Esophageal ulcer (Gastrointestinal disorders) | 0 | 1 — Adeers not subm
Esophagitis (Gastrointestinal disorders) | 0 | 2 — Adeers not subm
Eye disorders - Other, specify (Eye disorders) | 1 | 1 — Adeers not subm
Febrile neutropenia (Blood and lymphatic system disorders) | 29 | 20 — Adeers not subm
Fever (General disorders) | 6 | 2 — Adeers not subm
Fibrinogen decreased (Investigations) | 2 | 2 — Adeers not subm
Gastritis (Gastrointestinal disorders) | 1 | 0 — Adeers not subm
GGT increased (Investigations) | 3 | 0 — Adeers not subm
Headache (Nervous system disorders) | 16 | 4 — Adeers not subm
Hematoma (Vascular disorders) | 1 | 0 — Adeers not subm
Hematuria (Renal and urinary disorders) | 1 | 0 — Adeers not subm
Hepatic infection (Infections and infestations) | 0 | 1 — Adeers not subm
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 — Adeers not subm
Hyperglycemia (Metabolism and nutrition disorders) | 13 | 4 — Adeers not subm
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 1 — Adeers not subm
Hypernatremia (Metabolism and nutrition disorders) | 2 | 1 — Adeers not subm
Hypertension (Vascular disorders) | 3 | 2 — Adeers not subm
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 2 — Adeers not subm
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 2 — Adeers not subm
Hypokalemia (Metabolism and nutrition disorders) | 13 | 9 — Adeers not subm
Hyponatremia (Metabolism and nutrition disorders) | 4 | 2 — Adeers not subm
Hypophosphatemia (Metabolism and nutrition disorders) | 5 | 3 — Adeers not subm
Hypotension (Vascular disorders) | 4 | 5 — Adeers not subm
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 8 | 3 — Adeers not subm
Infections and infestations - Other, specify (Infections and infestations) | 15 | 15 — Adeers not subm
Insomnia (Psychiatric disorders) | 0 | 1 — Adeers not subm
Intracranial hemorrhage (Nervous system disorders) | 0 | 1 — Adeers not subm
Investigations - Other, specify (Investigations) | 0 | 1 — Adeers not subm
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Adeers not subm
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Adeers not subm
Lip infection (Infections and infestations) | 0 | 2 — Adeers not subm
Lipase increased (Investigations) | 1 | 0 — Adeers not subm
Lung infection (Infections and infestations) | 3 | 6 — Adeers not subm
Lymph gland infection (Infections and infestations) | 1 | 0 — Adeers not subm
Lymphocyte count decreased (Investigations) | 2 | 1 — Adeers not subm
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 | 0 — Adeers not subm
Mucosal infection (Infections and infestations) | 0 | 1 — Adeers not subm
Mucositis oral (Gastrointestinal disorders) | 12 | 7 — Adeers not subm
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 | 1 — Adeers not subm
Nail infection (Infections and infestations) | 1 | 0 — Adeers not subm
Nausea (Gastrointestinal disorders) | 6 | 0 — Adeers not subm
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — Adeers not subm
Nervous system disorders - Other, specify (Nervous system disorders) | 1 | 0 — Adeers not subm
Neutrophil count decreased (Investigations) | 4 | 2 — Adeers not subm
Oral hemorrhage (Gastrointestinal disorders) | 1 | 1 — Adeers not subm
Oral pain (Gastrointestinal disorders) | 3 | 2 — Adeers not subm
Otitis externa (Infections and infestations) | 1 | 0 — Adeers not subm
Otitis media (Infections and infestations) | 2 | 1 — Adeers not subm
Pain (General disorders) | 1 | 8 — Adeers not subm
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 — Adeers not subm
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 — Adeers not subm
Pancreatitis (Gastrointestinal disorders) | 3 | 0 — Adeers not subm
Papilledema (Eye disorders) | 0 | 1 — Adeers not subm
Papulopustular rash (Infections and infestations) | 1 | 0 — Adeers not subm
Pharyngitis (Infections and infestations) | 1 | 0 — Adeers not subm
Platelet count decreased (Investigations) | 3 | 0 — Adeers not subm
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3 — Adeers not subm
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Adeers not subm
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 — Adeers not subm
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 — Adeers not subm
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 3 — Adeers not subm
Rectal fistula (Gastrointestinal disorders) | 1 | 0 — Adeers not subm
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0 — Adeers not subm
Rectal pain (Gastrointestinal disorders) | 1 | 2 — Adeers not subm
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | 0 — Adeers not subm
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Adeers not subm
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 | 0 — Adeers not subm
Retinoic acid syndrome (Respiratory, thoracic and mediastinal disorders) | 4 | 1 — Adeers not subm
Retinopathy (Eye disorders) | 0 | 1 — Adeers not subm
Sepsis (Infections and infestations) | 1 | 0 — Adeers not subm
Sinusitis (Infections and infestations) | 2 | 1 — Adeers not subm
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 0 — Adeers not subm
Skin infection (Infections and infestations) | 5 | 1 — Adeers not subm
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1 — Adeers not subm
Small intestine infection (Infections and infestations) | 0 | 1 — Adeers not subm
Soft tissue infection (Infections and infestations) | 2 | 0 — Adeers not subm
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 2 — Adeers not subm
Splenic infection (Infections and infestations) | 0 | 1 — Adeers not subm
Stoma site infection (Infections and infestations) | 1 | 0 — Adeers not subm
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Adeers not subm
Suicide attempt (Psychiatric disorders) | 1 | 1 — Adeers not subm
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 | 0 — Adeers not subm
Thromboembolic event (Vascular disorders) | 3 | 1 — Adeers not subm
Tooth infection (Infections and infestations) | 0 | 1 — Adeers not subm
Toothache (Gastrointestinal disorders) | 1 | 0 — Adeers not subm
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Adeers not subm
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 | 1 — Adeers not subm
Typhlitis (Gastrointestinal disorders) | 2 | 1 — Adeers not subm
Upper respiratory infection (Infections and infestations) | 2 | 3 — Adeers not subm
Urinary tract infection (Infections and infestations) | 3 | 0 — Adeers not subm
Vaginal infection (Infections and infestations) | 1 | 0 — Adeers not subm
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1 — Adeers not subm
Ventricular arrhythmia (Cardiac disorders) | 1 | 1 — Adeers not subm
Ventricular tachycardia (Cardiac disorders) | 0 | 1 — Adeers not subm
Vitreous hemorrhage (Eye disorders) | 2 | 0 — Adeers not subm
Vomiting (Gastrointestinal disorders) | 6 | 0 — Adeers not subm
Vulval infection (Infections and infestations) | 1 | 0 — Adeers not subm
Weight gain (Investigations) | 1 | 0 — Adeers not subm
Weight loss (Investigations) | 3 | 0 — Adeers not subm
White blood cell decreased (Investigations) | 3 | 0 — Adeers not subm
Wound infection (Infections and infestations) | 2 | 0 — Adeers not subm

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.